CLINICAL TRIAL: NCT06062719
Title: Role of Octreotide Intravenous Infusion in Non-variceal GI Bleeding in ICU
Brief Title: Role of Octreotide in Non Variceal Bleeding
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Hepatology & Tropical Medicine Research Institute (Other Government)
Responsible Party: Principal Investigator, ICU, fellow of intensive care medicine, National Hepatology & Tropical Medicine Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 26-2023
Record Dates: First submitted 2023-08-29; First posted 2023-10-02 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Non-variceal Gastrointestinal Bleeding
MeSH Terms: interventions — Octreotide

STUDY DESIGN:
Intervention Model Description: Enrolled patients were assigned to one of two groups. After the initial endoscopy, both groups received either an 80-mg bolus of PPI alone (control group= A), followed by continuous intravenous (IV) infusion at 8 mg/h for a total of 72 hours or the octreotide adjunctive group, in addition to the pantoprazole (Study group= B) for 72 h, received a 100-μg bolus of octreotide, followed by continuous IV infusion of 50 μg/h for a total of 72 hours.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Active Comparator): 80-mg bolus of PPI alone (control group= A), followed by continuous intravenous (IV) infusion at 8 mg/h for a total of 72 hours
  Interventions: Drug: PPI group
- study (Experimental): octreotide adjunctive group, in addition to the pantoprazole (Study group= B) for 72 h, received a 100-μg bolus of octreotide, followed by continuous IV infusion of 50 μg/h for a total of 72 hours
  Interventions: Drug: PPI plus octreotide

INTERVENTIONS:
Drug: PPI group — 80-mg bolus of PPI alone (control group= A), followed by continuous intravenous (IV) infusion at 8 mg/h for a total of 72 hours
  Arms: control
Drug: PPI plus octreotide — octreotide adjunctive group, in addition to the pantoprazole (Study group= B) for 72 h, received a 100-μg bolus of octreotide, followed by continuous IV infusion of 50 μg/h for a total of 72 hours
  Arms: study

SUMMARY:
The rationale for using somatostatin (octreotide0 is that it has been shown to inhibit the secretion of various gastrointestinal hormones, including gastrin and secretin, which can contribute to the development of non-variceal gastrointestinal bleeding (NVGIB). Somatostatin has also been found to reduce splanchnic blood flow, which can decrease the risk of rebleeding in patients with NVGIB.

Previous studies have suggested that somatostatin may be effective in reducing the risk of rebleeding in patients with NVGIB, but there is a lack of high-quality randomized controlled trials evaluating its efficacy.

Therefore, this study aims to provide more rigorous evidence regarding the use of somatostatin in the management of NVGIB.

Aim of the study:

To evaluate the efficacy of medical treatment with somatostatin analogue (octreotide) combined with PPI in the treatment of non-variceal gastrointestinal bleeding in comparison to PPI alone a randomized.

DETAILED DESCRIPTION:
All patients admitted will receive the routine monitoring for the vital signs and supportive treatment. Resuscitation of a hemodynamically unstable patient begins with assessing and addressing the "ABCs" (i.e. airway, breathing, circulation) of initial management. Patients who are at an increased risk for aspiration, should be electively intubated. Intravenous access will be inserted and fluid resuscitation, blood, and blood products transfusion according to laboratory results. Nasogastric tune will be inserted andperform lavage, and endoscopic consultation post resuscitation within 24 hours.

Enrolled patients were assigned to one of two groups. After the initial endoscopy, both groups received either an 80-mg bolus of PPI alone (control group= A), followed by continuous intravenous (IV) infusion at 8 mg/h for a total of 72 hours or the octreotide adjunctive group, in addition to the pantoprazole (Study group= B) for 72 h, received a 100-μg bolus of octreotide, followed by continuous IV infusion of 50 μg/h for a total of 72 hours.

Hourly monitoring for vital signs including pulse, blood pressure, respiratory rate, oxygen saturation by pulse oximetry, 24hours urine output. Daily follow up for complete blood count, coagulation profile, urea, and creatinine will be done.

ELIGIBILITY:
Inclusion Criteria:

* The subjects are adults aged ≥18years old
* admitted to the intensive care unit of the National hepatology and Tropical Medicine Research institute and Alexandria university presenting with acute non-variceal gastrointestinal bleeding

Exclusion Criteria:

* If they have variceal bleeding
* received active endoscopic treatment (e.g. hemoclips or monopolar coagulation)
* known hypersensitivity to somatostatin analogue (octreotide) or any of its components
* pregnancy or breastfeeding
* active malignancy
* and use of somatostatin analogue within the past 7 day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-08-23 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
incidence of rebeeding | 7 days
  efficacy of octreotide infusion on the incidence of rebleeding7 days post randomization.

SECONDARY OUTCOMES:
blood transfusion | during 72 hours
  units of transfusions
length of stay | during the study UP TO 24 weeks
  ICU stay
length of stay | during the study up to 24 weeks
  hospital stay
mechanical ventilation | 72 hours
  incidence of need for mechanical ventilation
mortality | during the study up to 24 weeks
  non bleeding cause of mortality

CONTACTS AND LOCATIONS:
Locations (1):
- NHTMRI, Cairo, Egypt